CLINICAL TRIAL: NCT06462040
Title: Evaluation of Clinical and Radiological Outcomes in Patients Undergoing Fixation of Osteochondral Fragments With Reasorbable Screws in the Knee Joint
Acronym: OC-FIX
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: OC-FIX
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Osteochondral Defect; Osteochondritis Dissecans; Osteochondral Fracture; Osteochondral Fracture of Patella
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Fixation of osteochdral fragments with reabsorbable screws — Arthroscopic or mini-open fixation of free-intrarticular or unstable osteochondral fragments due to osteochondritis dissecans or osteochondral fractures with reabsorbable screws

SUMMARY:
Various techniques for the fixation of unstable osteochondral fragments have been used over the years, each with associated advantages and disadvantages, and differing clinical outcomes. However, the literature on the treatment of this type of injury in the adolescent and young adult population is scarce and involves small case series. Failure to treat these injuries can lead to serious consequences such as chronic pain, residual joint stiffness, and the development of early osteoarthritis, necessitating more invasive and burdensome interventions for the national health system, such as prosthetic replacements or osteotomies.

Due to the lack of real consensus within the scientific community regarding the ideal treatment for these patients and the insufficient medium/long-term follow-up data on the effects of these injuries on articular cartilage in young patients, this study aims to evaluate the clinical and radiological conditions of patients undergoing osteochondral fragment fixation using the same surgical technique (fixation with resorbable screws performed arthroscopically or via open surgery depending on the lesion's location) in order to clarify preventive measures against cartilage degeneration following these injuries, which are very common in adolescence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgical fixation of osteochondral fragment using resorbable screw technique, either arthroscopically or via mini-open procedure depending on the lesion's location, from 01/01/2017, and all new patients eligible for this type of intervention until 31/12/2025.
2. Patients aged between 12 and 35 years at the time of the surgical intervention.
3. Patients with the presence of osteochondral fragments confirmed by magnetic resonance imaging.
4. Patients with osteochondral lesions observed on imaging and symptoms attributable to the presence of osteochondral fragments.
5. Patients diagnosed with osteochondritis dissecans or recent contusion/sprain trauma.

Exclusion Criteria:

1. Patients with concomitant complex ligamentous injuries or fractures at the time of the intervention;
2. Patients who are no longer reachable;
3. Women of childbearing age who cannot exclude pregnancy;
4. Patients who are unable to provide informed consent or patients who are unwilling to sign the informed consent form.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from all subjects who have already undergone surgical treatment for fixation of knee osteochondral fragments using resorbable screws since 2017, and all new patients eligible for this type of intervention until 2025 at the Orthopedic and Traumatology Clinic II of the Rizzoli Orthopedic Institute.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
KOOS (Knee Injury and Ostearthritis Outcome Score) score | At least 24 months after surgery
  It represents a subjective score composed of 42 questions divided into 5 main domains. These domains investigate various aspects of symptoms and daily activities as well as the quality of life related to the knee and are divided as follows:
  * Symptoms, composed of 7 questions, 2 of which pertain to stiffness;
  * Pain, composed of 9 questions;
  * Functions and daily activities, composed of 17 questions;
  * Sports and recreational activities, composed of 5 questions;
  * Quality of life in relation to the knee, composed of 4 questions. All questions use the same response format, utilizing a quantitative scale ranging from 0 (no issues) to 4 (severe difficulty). Scores are calculated separately for each domain and converted into a percentage score, where 100 represents excellent physical condition with no symptoms and 0 represents severe disability with limitations in daily activities and constant symptoms even at rest.

SECONDARY OUTCOMES:
Kujala Anterior Knee Pain Scale | At least 24 months after surgery
  The Kujala score is a subjective knee assessment tool that quantifies limitations in daily and sports activities, as well as the presence or absence of symptoms. The questionnaire consists of 13 multiple-choice questions, with a total score ranging from 0 to 100. Each question has a variable score from 5 to 10 points and includes 3, 4, or 5 multiple-choice answers. The topics covered by each question include limping, pain, swelling, flexion deficit, and difficulty performing various types of activities. The maximum score of 100 represents no limitations or symptoms; the further the score deviates from 100, the worse the outcome.
International Knee Documentation Committee (IKDC) Score | At least 24 months after surgery
  The IKDC score is a subjective knee assessment tool that assesses limitations in daily and sports activities, as well as the presence or absence of symptoms.
  The IKDC score comprises three main domains:
  1. Symptoms, which include pain, stiffness, swelling, and the sensation of locking.
  2. Sports and daily activities.
  3. Current knee function and function before the injury.
  The questionnaire consists of 10 questions:
  * Seven items inquire about the patient's symptoms.
  * One item focuses on participation in sports.
  * One item, composed of 9 points, addresses the difficulties the patient experiences in performing daily activities.
  * The last item measures the current functionality of the knee.
  Scores range from 0 to 100, where 100 represents the absence of limitations and symptoms. The further the score deviates from 100, the worse the outcome, which can be categorized into four groups: excellent (80-100), good (60-80), fair (30-60), and poor (0-30).
Objective IKDC (IKDC standard evaluation form) | At least 24 months after surgery
  This represents a clinical chart that is completed by the physician following a comprehensive knee examination where various clinical tests are performed to assess for any joint deformities, objective instability, and meniscal injuries. The score obtained determines an objective evaluation grade coded using letters. According to this scale, grade "A" is assigned to a knee with "normal functionality, as healthy," grade "B" is assigned to a knee with "almost normal functionality," grade "C" is assigned to a knee with "moderately abnormal functionality," and grade "D" is assigned to a knee with "severely abnormal functionality."
MARX Activity Rating Scale | At least 24 months after surgery
  The MARX questionnaire is a subjective assessment tool designed to evaluate the activity level of patients with knee disorders who engage in sports. It focuses on four domains of sports activity: running, deceleration, cutting, pivoting.
  Patients are asked to approximate how many times they have performed each of these activities over the past twelve months. The four knee functions are evaluated on a 5-point frequency scale, and the scores are summed up to a maximum of sixteen points, where a higher score indicates more frequent participation and thus is correlated with a higher knee health status.
  The MARX questionnaire differs from many other activity measures because it is not based on participation in specific sports activities. Instead, patients are asked about different components of physical function (such as running and pivoting) common to various sports. The aim of this tool is to identify the overall activity level of the patient rather than their most recent activity.
VAS (Visual Analog Scale) for pain | At least 24 months after surgery
  This is a quantitative, one-dimensional numeric pain assessment scale, ranging from 0 to 10. The scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at the time of the visit and before the surgical intervention. 0 indicates no pain, while 10 indicates the worst possible pain.
Radiological evaluation (MRI, magnetic resonance imaging) throughout ICRS Cartilage Score | 24 months after surgery
  Assessment of healing of the fragment fixation
Radiological evaluation (MRI, magnetic resonance imaging) throughout Outerbridge Classification | 24 months after surgery
  Healing status of ostechondral fragment
Sports Activity Level, Tegner Score | At least 24 months after surgery
  Allows estimation of a subject's motor activity level with a score ranging from 0 to 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as national or international-level soccer. This score is commonly used to define the motor activity level of patients with knee disorders. Additionally, patients will be asked how many years they have been active in sports and whether the reduction or cessation of activity is related to knee pathology or not.
Thigh circumference | At least 24 months after surgery
  Measuring the circumference of the thigh at 5 cm and 15 cm from the superior pole of the patella allows for the evaluation of the degree of muscle trophism of the subjects under examination, and thus the potential influence of the type of technique used on muscle trophism.
Anterior knee pain / pain during knee flexion | At least 24 months after surgery
  In order to specifically assess the symptoms of the patellofemoral joint, patients will be asked to respond to these questions dichotomously (YES/NO).
Likert scale | At least 24 months after surgery
  In order to assess the level of patient satisfaction, they will be asked to respond to a question composed of 5 levels of satisfaction (from 1 to 5), where 1 indicates that the patient is very satisfied with the intervention, while 5 indicates a high degree of dissatisfaction.
Complications, subsequent interventions, or surgical failures | At least 24 months after surgery
  Any complications, subsequent interventions, and surgical failures will be documented and recorded in the CRF.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Rizzoli Orthopedic Institute, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
In the first phase, specialized medical personnel will identify eligible subjects within the hospital database. For retrospective cohorts, patients with provided contact details will be contacted, ensuring their consent for research participation. Interested patients will schedule a follow-up visit, during which they'll receive informational material and provide informed consent. Patients undergoing revision surgery or with septic arthritis will be considered surgical failures and excluded from follow-up. In the second phase, patients, after signing consent, will undergo clinical evaluation at least 24 months post-surgery, focusing on subjective assessments and clinical-instrumental tests. Knee MRI will evaluate radiological healing, with MRIs performed if documentation is unavailable. Visits will occur at the research clinic, and data will be recorded in Case Report Forms. The data will be entered into the RedCap Database.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code